CLINICAL TRIAL: NCT00994331
Title: Randomized Feasibility Study Comparing the Clinical Utility of the Stereotaxis Navigant™ Computed Tomography Angiography Importation and Co- Registration Feature, the NaviView™ Assisted Navigation Feature, and Standard Angiography
Brief Title: Stereotaxis Computed Tomography (CT) Co-Registration Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment.
Sponsor: Stereotaxis (Industry)
Responsible Party: Patricia Gipson, Stereotaxis, Inc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM-CLIN-011
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Magnetic Navigation; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A-CT Coregistration (Active Comparator): 5 subjects with CT co-registration in a magnetically navigated PCI (Group A)
  Interventions: Procedure: Percutaneous coronary intervention
- Group B-Angiographic (Active Comparator): 5 subjects with angiographic co-registration in a magnetically navigated PCI (Group B)
  Interventions: Procedure: Percutaneous coronary intervention
- Group C-Standard Angiography (Active Comparator): 5 subjects with standard angiography in a conventional PCI (Group C)
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — non surgical procedure to open blocked coronary arteries

SUMMARY:
The Stereotaxis Niobe® II Magnetic Navigation System (MNS) is designed to direct and digitally control catheter and guidewire based therapeutic and diagnostic devices along complex trajectories within the heart and coronary vasculature.

Navigation using vectors acquired from the CT Co-registration feature of Navigant™ provides clinical benefits for percutaneous coronary intervention (PCI) by decreasing the amount of contrast used during complex PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18-80 years of age
* Willing and able to provide prior written informed consent
* Patients present with a single bifurcated lesion or single non-CTO complex lesion requiring PCI.
* Able to be safely exposed to magnetic fields, such as magnetic resonance imaging (MRI)
* CT angiography performed prior to cardiac catheterization (must be performed >48 hours prior to procedure to limit peri-procedural contrast use, but <12 months prior to the procedure)

Exclusion Criteria:

* Patients with a creatinine greater than 2.0 mg/dL
* Exclude patients whom in the Investigator's opinion, are hemodynamically unstable on the day of the procedure.
* Untreatable allergy to contrast media
* Patients who have undergone CT angiography within 48 hours of index PCI procedure
* Patients with chronic total occlusions (CTOs) requiring intervention.
* Patients requiring treatment for lesions other than the single bifurcated or single non-CTO complex lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to compare and evaluate the total contrast use between Groups A, B and C . | 6 months

SECONDARY OUTCOMES:
The secondary endpoint is to compare and evaluate the following data points between Groups A, B and C: fluoroscopy time, procedure time, crossing time, procedural contrast use, adverse events (AEs): e.g. clinically significant perforations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Moses, MD, Principal Investigator — New York Presbyterian Hospital-Columbia Medical Center
Locations (1):
- New York Presbyterian Hospital-Columbia Medical Center, New York, New York, United States